CLINICAL TRIAL: NCT04067089
Title: Prospective, Randomized, Cost-utility Analysis of Transcatheter Aortic Valve Implantation Versus Surgical Aortic Valve Replacement in Brazil
Brief Title: Treatment of Aortic Stenosis in Brazil: Cost-Utility Analysis of TAVI vs SAVR
Acronym: TEAm-BR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hospital do Coracao (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TEAm-BR
Record Dates: First submitted 2019-08-11; First posted 2019-08-26 (Actual); Last update posted 2023-03-02 (Actual); Status verified 2023-03

CONDITIONS: Aortic Stenosis
Keywords: aortic stenosis
MeSH Terms: conditions — Aortic Valve Stenosis | interventions — Transcatheter Aortic Valve Replacement

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TAVR - Transcatheter aortic valve replacement (Experimental): TAVR - Transcatheter aortic valve replacement with Acurate Neo bioprosthesis (Boston Scientific) using minimalist approach
  Interventions: Procedure: TAVR - Transcatheter aortic valve replacement
- Surgical aortic valve replacement (Active Comparator): Surgical aortic valve replacement
  Interventions: Procedure: Surgical aortic valve replacement

INTERVENTIONS:
Procedure: TAVR - Transcatheter aortic valve replacement — TAVR - Transcatheter aortic valve replacement with Acurate Neo bioprosthesis (Boston Scientific) using minimalist approach
  Other Names: TAVR
  Arms: TAVR - Transcatheter aortic valve replacement
Procedure: Surgical aortic valve replacement — Surgical aortic valve replacement
  Other Names: SAVR
  Arms: Surgical aortic valve replacement

SUMMARY:
TEAM-Br is a randomized, prospective, cost-utility study comparing transcatheter aortic valve implantation (TAVI) versus surgical aortic vale replacement in Brazil.

The study is sponsored by the national Minister of Health, through PROADI-SUS (Programa de Apoio ao Desenvolvimento Institucional do SUS).

DETAILED DESCRIPTION:
Transcatheter aortic valve implantation has been shown to be non-inferior to surgical aortic valve replacement in patients with severe aortic stenosis at high, intermediate and low surgical risk. In recent years, a concept of a simplified and optimized TAVR procedure (known as minimalist approach) has led experienced centers to perform the majority of these procedures using conscious sedation and local anesthesia only. From a clinical perspective, this approach is associated with better and faster recovery and mobilization, reduced need for a prolonged intensive care unit (ICU) stay and faster hospital discharge, as compared to general anesthesia.

The cost-effectiveness of minimalist TAVR strategy - as compared to surgery - in Brazil is uncertain. Our objective is to conduct a cost-utility analysis comparing minimalist transcatheter aortic valve implantation with surgical aortic valve replacement in patients with severe aortic stenosis.

ELIGIBILITY:
Inclusion Criteria:

* Age > 70 years;
* Symptoms of heart failure NYHA class > II;
* Severe aortic stenosis (as defined by echocardiography: mean gradient >40 mmHg or jet velocity greater than 4.0 m/s or an initial aortic valve area of < 1.0 cm2)
* Heart team (including examining cardiac surgeon) agree on eligibility including assessment that TAVR or SAVR is appropriate;
* The study patient or the study patient's legal representative informed of the nature of the study, agreed to its provisions and provided written informed consent as approved by the Institutional Review Board (IRB) center;
* The study patient agreed to comply with all required post-procedure follow-up visits including visits through 1 month and 1 year;
* Heart team agreed (a priori) on treatment strategy for concomitant coronary disease (if present);
* Patient agreed to undergo surgical aortic valve replacement (SAVR) if randomized to control treatment.

Exclusion Criteria:

* Heart Team assessment of inoperability (including examining cardiac surgeon);
* Hostile chest
* Evidence of an acute myocardial infarction ≤ 1 month (30 days) before the intended treatment [defined as: Q wave MI, or non-Q wave MI with total CK elevation of CK-MB ≥ twice normal in the presence of MB elevation and/or troponin level elevation (WHO definition)];
* Concomitant severe valvular disease (mitral, tricuspid or pulmonic) requiring surgical intervention;
* Preexisting mechanical or bioprosthetic aortic valve with dysfunction;
* Complex coronary artery disease: unprotected left main coronary artery, Syntax score > 32 (in the absence of prior revascularization);
* Any therapeutic invasive cardiac procedure resulting in a permanent implant that is performed within 30 days of the index procedure (unless part of planned strategy for treatment of concomitant coronary artery disease). Implantation of a permanent pacemaker is not an exclusion criteria;
* Leukopenia (WBC < 3000 cell/mL), acute anemia (Hgb < 9 g/dL), thrombocytopenia (Plt < 50,000 cell/mL);
* Hypertrophic cardiomyopathy with or without obstruction (HOCM);
* Severe ventricular dysfunction with LVEF < 20%;
* Echocardiographic evidence of intracardiac mass, thrombus or vegetation;
* Active upper GI bleeding within 3 months (90 days) prior to procedure;
* A known contraindication or hypersensitivity to all anticoagulation regimens, or inability to be anticoagulated for the study procedure;
* Clinically (by neurologist) or neuroimaging confirmed stroke or transient ischemic attack (TIA) within 6 months (180 days) of the procedure;
* Renal insufficiency (creatinine > 3.0 mg/dL) and/or renal replacement therapy at the time of screening;
* Estimated life expectancy < 24 months (730 days) due to carcinomas, chronic liver disease, chronic renal disease or chronic end stage pulmonary disease;
* Currently participating in an investigational drug or another device study;
* Active bacterial endocarditis within 6 months (180 days) of procedure;
* Patient refuses surgery for aortic valve replacement.

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2018-12-10 (Actual); Primary Completion 2023-09-13 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Cost-utility of minimalist TAVR as compared to SAVR | 1 year
  Quality-adjusted life-years (QALYs). Quality of life will be assessed by EuroQol 5D.
Cost-utility of minimalist TAVR as compared to SAVR | 1 year
  Incremental cost-effectiveness ratio (ICER)

SECONDARY OUTCOMES:
Clinical outcomes | 30 days and 1 year
  All-cause mortality, cardiovascular mortality, disabling stroke, acute renal failure, bleeding, major vascular complications, atrial fibrillation and permanent pacemaker implantation

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre A Abizaid, MD, PhD, Study Chair — Hospital do Coracao; Fabio Jatene, MD, PhD, Study Chair — Hospital do Coracao; Dimytri A Siqueira, MD PhD, Principal Investigator — Hospital do Coracao; Paulo P Fernandes, Md, PhD, Study Chair — Hospital do Coracao
Locations (1):
- Hospital do Coracao, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
Reproducible Research Statement:We will share the database containing de-identified individual participant data, data dictionary documentation, statistical analysis plan, and analysis code.
  Beginning 6 months and ending 24 months following article publication, the trial steering committee will evaluate proposals of studies accompanied by a statistical analysis plan and may grant access to the data for approved proposals. After 24 months, the database and accompanying documents will be publicly available in an institutional data repository (http://www.hcor.com.br).
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Beginning 6 months and ending 24 months following article publication, the trial steering committee will evaluate proposals of studies accompanied by a statistical analysis plan and may grant access to the data for approved proposals. After 24 months, the database and accompanying documents will be publicly available in an institutional data repository (http://www.hcor.com.br).
URL: http://www.hcor.com.br